CLINICAL TRIAL: NCT04143295
Title: Rescue of Infants With MCT8 Deficiency
Acronym: DITPA
Status: Available | Type: Expanded Access
Sponsor: Roy E. Weiss, M.D. (Other)
Responsible Party: Sponsor-Investigator, Roy E. Weiss, M.D., Principal Investigator, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20180087
Record Dates: First submitted 2018-04-24; First posted 2019-10-29 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Mct8 (Slc16A2)-Specific Thyroid Hormone Cell Transporter Deficiency
MeSH Terms: conditions — Allan-Herndon-Dudley syndrome | interventions — 3,5-diiodothyropropionic acid

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Diiodothyropropionic acid (DITPA) — Drug Administration

SUMMARY:
Monocarboxylate Transporter 8 (MCT8) deficiency (that is also known as Allan-Herndon-Dudley syndrome) is a rare X-linked inherited disorder of brain development that causes severe intellectual disability and problems with movement. This condition, which occurs almost exclusively in males, disrupts development from before birth.

ELIGIBILITY:
Inclusion Criteria

* Genetic Confirmation: Male fetus or fetuses (including monozygotic twin pregnancies) must have a confirmed MCT8 gene mutation.
* Family History: A previously born child or children with a severe, typical phenotype and an MCT8 gene mutation identical to that of the fetus.
* Alternatively, the mother or a sister must have a relative with a known MCT8 defect.
* Parental Decision: Parental refusal to terminate the pregnancy despite the diagnosis of MCT8 deficiency.
* Compliance and Availability: Willingness of the parents to comply with all study procedures and ensure availability for the duration of the study.

Exclusion Criteria:

• Pregnancy-Related Factors: Dizygotic (non-identical) twin pregnancy (unless only one fetus is confirmed with the MCT8 mutation, and the unaffected fetus will not be treated).

Parental decision to terminate the pregnancy.

• Maternal Medical Conditions: Hyperthyroidism requiring treatment. Significant liver or kidney insufficiency. Congestive heart failure. Hyperemesis gravidarum unresponsive to treatment.

* Significant cardiac conditions, including:
* Atrial fibrillation or other arrhythmias.
* Unstable angina.
* Coronary heart disease.
* Medications:

Current use of sympathomimetic therapy. Anticoagulant therapy. Use of Cytochrome P450 2C9 (CYP2C9) inhibitors with a narrow therapeutic index.

• Other Factors: Major illness or recent major surgery within four weeks of baseline visit 1, unrelated to MCT8 deficiency.

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — MCT8 mutation carrier mother with previously affected MCT8 deficient male will be screened for male fetal DNA as soon as she aware she is pregnant (week 4-7).

CONTACTS AND LOCATIONS:
Overall Officials: Roy E Weiss, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miller School of Medicine, Miami, Florida, United States